CLINICAL TRIAL: NCT07314411
Title: Effect of Carotenoid Supplementation on Retinal Health: An Evaluation of Macular Structure and Function in Healthy Adults
Brief Title: Carotenoid Supplementation and Retinal Health in Healthy Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pacific University (Other)
Collaborators: MacuHealth (Industry)
Responsible Party: Principal Investigator, Aditi Deshpande, Principal Investigator, Pacific University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: IRB 132-24
Record Dates: First submitted 2025-12-05; First posted 2026-01-02 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment- Carotenoid Supplementation (Experimental)
  Interventions: Dietary Supplement: other
- Placebo (Experimental)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: other — Participant will be provided with a commercially-made softgel capsule (either carotenoid supplement or placebo containing only the inactive ingredients) in unmarked bottles and instructed to take one softgel capsule daily with a meal for 3 months.
  Arms: Treatment- Carotenoid Supplementation
Dietary Supplement: Placebo — Participant will be provided with a commercially-made softgel capsule (either carotenoid supplement or placebo containing only the inactive ingredients) in unmarked bottles and instructed to take one softgel capsule daily with a meal for 3 months.
  Arms: Placebo

SUMMARY:
The purpose of this research is to evaluate the effect of oral dietary carotenoid supplements on various aspects of retinal health. This includes assessing its impact on macular pigment optical density (MPOD), which is a protective feature of retinal health in reducing lipofuscin (retinal waste) accumulation in the retina.

Our goal is to investigate the protective role of this oral carotenoid supplement on the macular structure, measured as retinal thickness, macular blood vessel density, choriocapillaris density and ocular perfusion pressure (defined as the difference between blood pressure and eye pressure) as well as evaluating visual functions such as contrast sensitivity (the ability to perceive less bold objects ) and photostress recovery time (the minimum time for a person to read the lowest level on an eye chart after shining a light in front of the eye for several seconds). This study will also investigate the relationship between skin carotenoid level and ocular carotenoid level, using a non-invasive finger measurement. Also, we want to explore the effect of carotenoid supplementation on cognitive function in terms of working memory. Understanding how this supplementation impacts all these markers is crucial for enhancing our knowledge of the potential health benefits of carotenoids in improving dietary assessment methods.

This study takes 3 visits. Participants will provide written informed consent on the first visit after reviewing the study procedures, potential risks, benefits, confidentiality measures, and their right to withdraw. Then they will undergo a comprehensive history-taking and complete a validated questionnaire to screen for sensitivity to light, as well as a diet questionnaire. Following this, participant will have non-invasive testing, requiring no eye drops or dyes. This involves measurement of contrast sensitivity (CS), photostress recovery, MPOD, blood pressure (BP), intraocular pressure (IOP), skin carotenoid level, retinal thickness and vascular measures using an optical coherence tomographer (OCT), lipofuscin levels using fundus autofluorescence (FAF) pictures and cognitive function assessment of working memory using a computerized 2- back test. Each participant will then be provided with a commercially-made softgel capsule (either carotenoid supplement or placebo containing only the inactive ingredients) in unmarked bottles and instructed to take one softgel capsule daily with a meal for 3 months. Follow-up visits will take place for 1 month and 3 months, during which the same measurements mentioned above will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-75 years
* Monocular best corrected visual acuity (BCVA) of 20/20 or better
* Eye pressure between 8 and 22 mm of Hg (will be screened in study if needed)
* Ability to provide informed consent
* Access to the Internet

Exclusion Criteria:

* History of or currently active eye diseases or systemic disease
* History of refractive surgery or ocular surgery
* Currently pregnant, nursing or planning to become pregnant during the study period
* Known allergy to any study active or inactive ingredient
* Current supplementation with any components of MacuHealth or placebo softgel capsules
* Drugs that may interact with absorption of fat-soluble vitamins/carotenoids especially orlistat and bile acid sequestrants (i.e., colestyramine, fat-free substitutes such as Olestra, beta-carotene, and vitamin E), or antidiabetic drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Macular Pigment Optical Density (MPOD) in Density Units Over 3 Months | From enrollment to the end of treatment at 3 months
Change From Baseline in Fundus Autofluorescence (FAF) Brightness in Pixels Over 3 Months | From enrollment to the end of treatment at 3 months

SECONDARY OUTCOMES:
Change From Baseline in Central Retinal Thickness in Micrometers (µm) Over 3 Months | From enrollment to the end of treatment at 3 months
Change From Baseline in Macular Vascular and Choriocapillaris Density in Percentage (%) Over 3 Months | From enrollment to the end of treatment at 3 months
Change From Baseline in Skin Carotenoid Levels measured as Score Over 3 Months | From enrollment to the end of treatment at 3 months
Change From Baseline in Memory Test Measured as Percentage (%) of Correct Responses Over 3 Months | From enrollment to the end of treatment at 3 months

OTHER OUTCOMES:
Change From Baseline in Contrast Sensitivity in Log Contrast Units Over 3 Months | From enrollment to the end of treatment at 3 months
Change From Baseline in Photostress Recovery Time (PRT) Measured in Seconds Over 3 Months | From enrollment to the end of treatment at 3 months
Change From Baseline in Mean Ocular Perfusion Pressure (OPP) Measured in Millimeters of Mercury (mmHg) Over 3 Months | From enrollment to the end of treatment at 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Pacific University, Forest Grove, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared at this time due to ongoing analyses.

REFERENCES:
- See also: The web page compiles information on scientific and clinical studies related to macular carotenoid supplements, nutrition, retinal health, and eye function. — https://www.macuhealth.com/learning-center/topic/learning-center-clinical-studies/